CLINICAL TRIAL: NCT01173328
Title: Effects of Pursed-lip Breathing on Exercise Tolerance and Dynamic Hyperinflation in Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Pursed-lip Breathing on Exercise Tolerance and Dynamic Hyperinflation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Leandro Ferracini Cabral, Universidade Federal de Juiz de Fora
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CEP/HUCFF/UFRJ 187/07
Record Dates: First submitted 2010-07-19; First posted 2010-08-02 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2008-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: exercise tolerance; dynamic hyperinflation; respiratory mechanics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pursed-lip Breathing (Experimental)
  Interventions: Behavioral: Pursed-lip breathing; Behavioral: Normal Breathing

INTERVENTIONS:
Behavioral: Pursed-lip breathing — Pursed-lip breathing involves a nasal inspiration followed by expiratory blowing against partially closed lips, avoiding forceful exhalation.
Behavioral: Normal Breathing

SUMMARY:
Pursed-lip breathing (PLB) has been advocated to reduce respiratory rate and improve oxygen saturation in patients with chronic obstructive pulmonary disease (COPD) at rest. Although PLB is a strategy that potentially reduces expiratory flow limitation, there are only few studies addressing its effects on exercise.

This study aimed to assess the ability of PLB to change the breathing pattern, degree of dynamic hyperinflation (DH) and arterial oxygenation in COPD patients during exercise. Exercise tolerance was evaluated by endurance time and respiratory mechanics was evaluated by forced oscillation technique.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease (COPD)
* Regular treatment at Clementino Fraga Filho University Hospital (UFRJ)

Exclusion Criteria:

* Exacerbation in the preceding 4 weeks
* SpO2<85% at peak exercise
* Other diseases that may contribute to dyspnea and exercise intolerance

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Endurance time | within the first 01 hour

SECONDARY OUTCOMES:
inspiratory capacity | within the first 01 hour
oxygen saturation | within the first 01 hour
dyspnea | within the first 01 hour
forced oscillation variables | within the first 01 hour

CONTACTS AND LOCATIONS:
Overall Officials: Fernando S Guimarães, PhD, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Clementino Fraga Filho University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil